CLINICAL TRIAL: NCT04701138
Title: Bioavailability of Specialized Pro-resolving Mediators in Obese Humans
Brief Title: Bioavailability of SPMs in Obese Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Metagenics, Inc. (Industry); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-0131; 550KR242033 (Other Grant/Funding Number: NC TraCS)
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Results first posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-03

CONDITIONS: Obesity Adult Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Supplement (Experimental): All subjects will receive the intervention (SPM Active Supplement)
  Interventions: Dietary Supplement: SPM Active

INTERVENTIONS:
Dietary Supplement: SPM Active — Each capsule contains 145 mg of SPMs (fractionated marine lipids standardized to 18-HEPE, 14-HDHA, and 17-HDHA). All subjects will take 4 capsules orally each day for a total daily dose of 580 mg.

SUMMARY:
Research Question: Does 4 weeks of supplementation with 'SPM Active' lead to a statistically significant increase in plasma SPM concentration for obese human subjects? Primary Aim 1: To compare plasma SPM concentrations and immunological fitness pre- and post- oral SPM administration in the obese.

* Aim 1a: To quantify plasma SPM concentrations in plasma (pg/mL), serum (pg/mL) and PBMCs before and after 4 weeks of supplementation with 'SPM Active.' The concentration of SPMs in plasma, in addition to other PUFA-derived metabolites that share the same enzymatic pathways as SPMs, will be established at baseline and post-intervention using mass spectrometry-based metabololipidomics.
* Aim 1b: To measure in vitro antibody responses of B cells in PBMC pool with in vitro stimulation and cytokine production before and after 4 weeks of supplementation with 'SPM Active.' In addition, researchers will quantify the relative abundance of differing immune cell populations.

DETAILED DESCRIPTION:
Purpose: Specialized pro-resolving mediators (SPMs) are a superfamily of lipid metabolites, predominantly derived from the n-3 polyunsaturated fatty acids (PUFAs) eicosapentaenoic (EPA) and docosahexaenoic acids (DHA). Previous research has established that obese mice and humans have lower circulating levels of SPMs relative to lean controls. In this study, SPMs will be administered as a dietary supplement to obese human subjects to establish: 1) their bioavailability in plasma, serum and peripheral blood mononuclear cells (PBMCs) and 2) their effects on immune cell abundance and in vitro antibody production. The rationale for focusing on immune cells is that SPMs may be targeting their abundance and phenotype. This study does not intend to make any health or health-related claims.

Participants: A total of 24 (n=12 men + 12 women) obese (BMI 30-40 kg/m2) euglycemic and pre-diabetic subjects (fasting glucose 70-125 mg/dL or HbA1c of 5.7-6.4%) aged 50-65 years will be recruited by Dr. Erik Butler from the UNC Family Medicine Center in Chapel Hill.

Procedures (methods): This is a non-randomized uncontrolled clinical trial. The study will provide the intervention 'SPM Active' provided by Metagenics. All subjects will be advised to take 4 capsules per day (2 capsules with breakfast and 2 capsules with dinner) of 'SPM Active' for 4 weeks total. Each capsule contains 145 mg of SPMs for a total daily dose of 580 mg. Fasting blood will be drawn pre- and post-intervention using phlebotomy available under the direction of Dr. Butler. The scientific approach will rely on mass-spectrometry based metabololipidomics, immunophenotyping with flow cytometry, and anthropomorphic/blood pressure/BMI measurements (anthropometric measures are only intended for use in statistical analysis for confounding variables).

ELIGIBILITY:
Inclusion Criteria:

* 24 (n=12 male + 12 female) obese (BMI 30-40 kg/m^2) subjects with age 50-65 years who are euglycemic and pre-diabetic (i.e. fasting glucose 70-125 mg/dL or HbA1c of 5.7-6.4%).
* Only post-menopausal females will be recruited in the female cohort to reduce the confounding effects of estrogen on lipid metabolism during supplementation.

Exclusion Criteria:

* Those with fasting glucose values > 126 mg/dL or known type 2 diabetes
* Females who are pre-menopausal, pregnant, planning to become pregnant, breastfeeding or lactating
* Subjects consuming n-3 PUFA supplements in the last 3 months prior to enrollment, high consumption of fatty fish (>2 servings per week), and subjects with active autoimmune disease, liver disease, coagulopathy, hypothyroidism, known allergy to fish or shellfish, inability to give informed consent, or taking anticoagulants (e.g. warfarin and direct-acting anticoagulants), those taking estrogen or testosterone, and anyone taking daily aspirin, NSAIDs, or active asthma medications.
* Subjects receiving immunomodulatory or immunosuppressant therapy (corticosteroids or monoclonal antibodies) in the 4 weeks prior to study enrollment, and subjects with known active malignancy or undergoing treatment for malignancy will be excluded.
* Subjects who test positive for COVID-19 or have tested positive in the past will be excluded. Those who report COVID-19 or flu-like symptoms will be excluded, as well as those that fail to pass COVID-19 screening at baseline.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saame R Shaikh, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Erik Butler, DO, Study Director — UNC Family Medicine
Locations (1):
- UNC Chapel Hill Family Medicine Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Each participant's deidentified metabololipidomics data and flow cytometry/immunophenotyping data will be shared via ImmPort
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available 24-36 months after the completion of the study. Data will be available permanently.
Access Criteria: Flow cytometry data will be deposited into ImmPort (https://www.immport.org/home). The raw metabololipidomics data will be made available by depositing the results in http://www.metabolomicsworkbench.org/. Analytic code and statistical analysis plans will be deposited on github.com. The study protocol, statistical analysis plan, & informed consent form will be made available on clinicaltrials.gov.

REFERENCES:
- [Background] Crouch MJ, Kosaraju R, Guesdon W, Armstrong M, Reisdorph N, Jain R, Fenton J, Shaikh SR. Frontline Science: A reduction in DHA-derived mediators in male obesity contributes toward defects in select B cell subsets and circulating antibody. J Leukoc Biol. 2019 Aug;106(2):241-257. doi: 10.1002/JLB.3HI1017-405RR. Epub 2018 Dec 21. PMID 30576001
- [Background] Kosaraju R, Guesdon W, Crouch MJ, Teague HL, Sullivan EM, Karlsson EA, Schultz-Cherry S, Gowdy K, Bridges LC, Reese LR, Neufer PD, Armstrong M, Reisdorph N, Milner JJ, Beck M, Shaikh SR. B Cell Activity Is Impaired in Human and Mouse Obesity and Is Responsive to an Essential Fatty Acid upon Murine Influenza Infection. J Immunol. 2017 Jun 15;198(12):4738-4752. doi: 10.4049/jimmunol.1601031. Epub 2017 May 12. PMID 28500069
- [Background] Serhan CN, Levy BD. Resolvins in inflammation: emergence of the pro-resolving superfamily of mediators. J Clin Invest. 2018 Jul 2;128(7):2657-2669. doi: 10.1172/JCI97943. Epub 2018 May 14. PMID 29757195
- [Background] Lopez-Vicario C, Titos E, Walker ME, Alcaraz-Quiles J, Casulleras M, Duran-Guell M, Flores-Costa R, Perez-Romero N, Forne M, Dalli J, Claria J. Leukocytes from obese individuals exhibit an impaired SPM signature. FASEB J. 2019 Jun;33(6):7072-7083. doi: 10.1096/fj.201802587R. Epub 2019 Mar 6. PMID 30840838
- [Derived] Al-Shaer AE, Regan J, Buddenbaum N, Tharwani S, Drawdy C, Behee M, Sergin S, Fenton JI, Maddipati KR, Kane S, Butler E, Shaikh SR. Enriched Marine Oil Supplement Increases Specific Plasma Specialized Pro-Resolving Mediators in Adults with Obesity. J Nutr. 2022 Jul 6;152(7):1783-1791. doi: 10.1093/jn/nxac075. PMID 35349683

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dietary Supplement
Started | 24
Completed | 23
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dietary Supplement
Number analyzed (Participants) | 23
Age, Continuous [Mean (Full Range); unit: years] | 56 [52 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
Weight [Median (Full Range); unit: Kg] | 96.4 [87.3 to 112.0]
Height [Median (Full Range); unit: cm] | 170.2 [160.0 to 177.8]
Body Mass Index (BMI) [Median (Full Range); unit: Kg/m^2] | 33.1 [31.0 to 36.0]

OUTCOME MEASURES:

1. Primary Outcome: Mean Pro-inflammatory & Pro-resolving Metabolites
Description: Mass spectrometry metabololipidomics analysis will be performed on plasma samples from pre/post supplementation blood draws to measure SPM concentrations. The study was powered to measure the following molecules of interest: 14-HDHA, 17-HDHA, and 18-HEPE.
Time Frame: From Baseline (Week 1/Day1) through 28 to 30 days of supplementation
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dietary Supplement
Number analyzed (Participants) | 23
ng/mL
  Pre 14-HDHA | 15.6 (11.5)
  Post 14-HDHA | 12.2 (5.4)
  Pre 17-HDHA | 6.6 (4.9)
  Post 17-HDHA | 8.1 (4.6)
  Pre 18-HEPE | 8.0 (6.2)
  Post 18-HEPE | 11.3 (10.3)

2. Secondary Outcome: Mean White Blood Cell Populations
Description: Immunological phenotyping of blood peripheral mononuclear cells (PBMC) using flow cytometry will identify key immune cell populations pre/post supplementation. PBMC analyses represent B cell populations, monocyte populations, natural killer cell populations, and T cell populations. The relative abundance was calculated using two different flow cytometry panels with fluorescently labeled antibodies. The first panel measured the relative abundance of all B cell subsets, monocyte subsets, and NK cell subsets (i.e., all subsets within error add up to 1.0). The second panel measured the relative abundance of CD4 T cell subsets, CD8 T cell subsets, and NKT cells (i.e., all subsets within error add up to 1.0).
Time Frame: From Baseline (Week 1/Day1) through 28 to 30 days of supplementation
Measure: Mean (Standard Deviation); unit: Relative abundance
Arm/Group | Dietary Supplement
Number analyzed (Participants) | 23
Relative abundance
  Pre CD4+ T Cells | 0.32 (0.07)
  Post CD4+ T Cells | 0.33 (0.05)
  Pre Activated CD4+ T Cells | 0.02 (0.01)
  Post Activated CD4+ T Cells | 0.03 (0.01)
  Pre Non-Activated CD4+ T Cells | 0.30 (0.07)
  Post Non-Activated CD4+ T Cells | 0.30 (0.05)
  Pre CD8 T Cells | 0.17 (0.07)
  Post CD8 T Cells | 0.16 (0.05)
  Pre Activated CD8 T Cells | 0.02 (0.01)
  Post Activated CD8 T Cells | 0.03 (0.02)
  Pre Non-Activated CD8 T Cells | 0.15 (0.06)
  Post Non-Activated CD8 T Cells | 0.13 (0.03)
  Pre NKT Cells | 0.02 (0.01)
  Post NKT Cells | 0.02 (0.01)
  Pre B Cells | 0.39 (0.08)
  Post B Cells | 0.37 (0.11)
  Pre Plasma Cells | 0.02 (0.01)
  Post Plasma Cells | 0.02 (0.01)
  Pre Follicular B Cells | 0.01 (0.01)
  Post Follicular B Cells | 0.01 (0.00)
  Pre B Regs | 0.08 (0.04)
  Post B Regs | 0.07 (0.04)
  Pre Classical Monocytes | 0.06 (0.02)
  Post Classical Monocytes | 0.06 (0.03)
  Pre Intermediate Monocytes | 0.00 (0.00)
  Post Intermediate Monocytes | 0.01 (0.00)
  Pre Non-Classical Monocytes | 0.11 (0.06)
  Post Non-Classical Monocytes | 0.10 (0.07)
  Pre NK CD3-CD56HICD16- | 0.01 (0.00)
  Post NK CD3-CD56HICD16- | 0.02 (0.03)
  Pre NK CD3-CD56HICD16+ | 0.01 (0.01)
  Post NK CD3-CD56HICD16+ | 0.02 (0.01)
  Pre NK CD3-CD56dimCD16- | 0.23 (0.09)
  Post NK CD3-CD56dimCD16- | 0.22 (0.08)
  Pre NK CD3-CD56dimCD16+ | 0.02 (0.01)
  Post NK CD3-CD56dimCD16+ | 0.02 (0.01)
  Pre NK CD3-CD56-CD16+ | 0.05 (0.03)
  Post NK CD3-CD56-CD16+ | 0.08 (0.08)

3. Other Pre Specified Outcome: Antibody Concentrations in Culture
Description: B cells isolated from collected blood samples will be cultured in-vitro and stimulated with an antigen & produced antibody concentrations will be measured via ELISA. This will be done for pre & post blood samples.
Time Frame: From Baseline (Week 1/Day1) through 28 to 30 days of supplementation
Population: One participant's sample was removed from all B cell isolation and stimulation studies (ELISA data) due to PBMC cell death upon sample freezing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dietary Supplement
Number analyzed (Participants) | 22
ng/mL
  Pre IgM | 465801.89 (217732.43)
  Post IgM | 457833.05 (238874.79)
  Pre IgG | 1024891.3 (394612.17)
  Post IgG | 789525.69 (320595.08)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through the last blood draw, ranging from 28 to 30 days.
Arm/Group | Dietary Supplement
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT04701138/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT04701138/ICF_001.pdf